CLINICAL TRIAL: NCT05786612
Title: A Randomised Controlled Investigation Comparing the Clinical Performance and Cost Effectiveness of Biatain® Silicone With Standard of Care Dressing Including Filler in Chronic Wounds
Brief Title: Clinical Performance and Cost Effectiveness of Biatain® Silicone Compared With Standard of Care
Acronym: BISIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP351
Record Dates: First submitted 2023-01-18; First posted 2023-03-27 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Venous Leg Ulcer; Diabetic Foot Ulcer
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The clinical investigation is a two-arms, open-labelled, stratified, randomized, controlled, multicentre investigation comparing the clinical performance of Biatain® Silicone with standard of care in chronic wounds with wound depth down to 20 mm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mepilex Border with Aquacel Extra Hydrofiber (Active Comparator): Standard of care (filler, that functions as a primary dressing to manage exudate and the gap/space between the wound bed and the dressing, covered by a secondary dressing on top) defined in this study as Mepilex® Border with AQUACEL® Extra Hydrofiber Dressing
  Interventions: Device: Mepilex Border with Aquacel Extra Hydrofiber
- Biatain® Silicone (Experimental): The investigational test product is Biatain® Silicone. Biatain® Silicone is intended to be used for moist wound healing and exudate management and can be used without a filler.
  Interventions: Device: Biatain® Silicone

INTERVENTIONS:
Device: Biatain® Silicone — Wound care dressing
  Arms: Biatain® Silicone
Device: Mepilex Border with Aquacel Extra Hydrofiber — Wound care dressing
  Arms: Mepilex Border with Aquacel Extra Hydrofiber

SUMMARY:
A randomised controlled investigation comparing the clinical performance and cost effectiveness of Biatain® Silicone with Standard of Care dressing including filler in chronic wounds (CP351 - BISIL Study)

This study (BISIL) will compare the Biatain® Silicone dressing to commonly used wound care products (AQUACEL®EXTRATM Hydrofiber® Dressing used with Mepilex® Border).

The study will recruit in total 100 adult subjects with a venous leg ulcer or a diabetic foot ulcer no deeper than 2cm. Only ulcers with a duration of at least 8 weeks but no longer than a year will be included. The study will be a randomised controlled trial where half of the participants will use Biatain® Silicone and half will use the comparator for 4 weeks. Each participant will be in the study for 4-5 weeks during which there will be a weekly visit with the study team to complete the study assessments and change the dressing. The study will run for approximately one year, starting in January 2023.

DETAILED DESCRIPTION:
A randomised controlled investigation comparing the clinical performance and cost effectiveness of Biatain® Silicone with Standard of Care dressing including filler in chronic wounds (CP351 - BISIL Study)

The properties of a wound dressing can have a significant impact on wound healing and on the risk of developing infections. The ideal wound dressing should have good contact with the wound and be effective in absorbing and holding fluids. Biatain® Silicone uses 3DFit technology, which may support better contact with the wound, help to absorb fluid more effectively and reduce the risk of leakage. These properties may support faster wound healing and reduce complications.

This study (BISIL) will compare the Biatain® Silicone dressing to commonly used wound care products (AQUACEL®EXTRATM Hydrofiber® Dressing used with Mepilex® Border). All products used in this study are CE-marked medical devices which are already available in the UK. The main objective is to compare the reduction in wound area over four weeks between the two treatment groups. The study will also look at other aspects of wound healing and compare the costs of the dressings and the participants' quality of life during the study period. In a subgroup of participants, ultrasound will be used to assess the contact between the dressings and the wound.

The study will recruit in total 100 adult subjects with a venous leg ulcer or a diabetic foot ulcer no deeper than 2cm. Only ulcers with a duration of at least 8 weeks but no longer than a year will be included. Participants will be inpatients or outpatients recruited through 12-18 Tissue Viability Units and hospitals across the UK. The study will be a randomised controlled trial where half of the participants will use Biatain® Silicone and half will use the comparator for 4 weeks. Each participant will be in the study for 4-5 weeks during which there will be a weekly visit with the study team to complete the study assessments and change the dressing. The study will run for approximately one year, starting in January 2023.

ELIGIBILITY:
Inclusion Criteria:

* Has given written consent to participate by signing the Informed Consent Signature Form
* Is at least 18 years of age and has full legal capacity
* Has a venous leg ulcer (VLU) (C6 of the CEAP classification(1)) or a non-infected diabetic foot ulcer (DFU) with a duration longer than 8 weeks but no longer than 24 months
* Has a wound with depth1 down to 20 mm
* Has a maximum wound depth1 relative to wound diameter
* Has a wound with exudate levels requiring a filler and a standard secondary dressing
* Has acceptance of compression therapy in case of a VLU or off-loading in case of a DFU, according to local standards
* For subjects with diabetes, has HbA1c ≤ 10% or ≤ 86 mmol/mol, measured within the last 3 months prior to inclusion

Exclusion Criteria:

* Wound is infected. For DFUs, has infection severity mild-severe according to the IWGDF/IDSA guideline For VLUs, has 2 or more clinical signs of infection as defined in protocol, based on clinical judgement by investigator/tissue viability nurse
* Wounds is with exposed tendons, is with bones or has fistulas
* Wound is with cavity, or is undermined or tunnelling
* Subject is receiving chemotherapy
* Subject has ankle-brachial pressure index (ABPI) below 0.8 measured within one month prior to inclusion
* Wound is larger than 10 x10 cm
* Currently enrolled in another wound care de-vice investigation unless co-enrolment has been agreed with the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Voegeli, Study Chair — University of Winchester
Locations (9):
- United Kingdom (9):
  - Norfolk Community Health and Care NHS Trust, Norwich, Bowthorpe Road Norwich
  - Milton Keynes University Hospital, Milton Keynes, Buckinghamshire
  - North Cumbria Integrated Care, Carlisle, Cumbria
  - Homerton Hospital, London, Greater London
  - Somerset NHS Foundation Trust, Taunton, Somerset
  - Torbay and South Devon, Torquay, Torbay
  - Leeds Teaching Hospitals, Leeds, West Yorkshire
  - Northumbria Healthcare, Ashington
  - Pioneer Wound care and Lymphoedema Centres, Eastbourne

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mepilex Border With Aquacel Extra Hydrofiber | Biatain® Silicone
Started | 51 | 51
Completed | 50 | 47
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 2
Not completed — one screening failure | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants included subjects with chronic wounds up to 2cm of depths with either venous leg ulcers or diabetic foot ulcers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mepilex Border With Aquacel Extra Hydrofiber | Biatain® Silicone | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (12) | 69.7 (12) | 71.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 28 | 30 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (9.6) | 30.4 (7.8) | 30.4 (8.7)
Wound type: Venous leg ulcer; diabetic foot ulcer [Count of Participants; unit: Participants]
  Venous leg ulcer | 40 | 39 | 79
  Diabetic foot ulcer | 11 | 12 | 23
Wound age (month) [Mean (Standard Deviation); unit: months] | 5.7 (4.8) | 5.1 (4.4) | 5.4 (4.6)
Wound depth (mm) [Mean (Standard Deviation); unit: mm] | 2.7 (2.3) | 2.3 (2) | 2.5 (2.2)
Wound area (subtracted islands) (cm2) [Mean (Standard Deviation); unit: cm2] | 5.6 (6.1) | 6.1 (8.8) | 5.8 (7.5)
Comorbidities [Count of Participants; unit: Participants]
  Diabetes | 16 | 16 | 32
  Venous insufficiency | 43 | 41 | 84
  Peripheral arterial disease | 8 | 5 | 13
  Cardiopulmonary conditions | 13 | 19 | 32
  Immune deficiencies | 3 | 2 | 5
  Other | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage Wound Area Reduction (WAR) During Four Weeks
Description: Photos of the wounds were collected at every site visit. A ruler or marker was used for calibration of linear dimensions at the image. Wound size reduction between visit 5 and at baseline was calculated. The mean WAR for each treatment group was calculated. As wounds would become smaller over time, the baseline wound size minus the wound size at visit 5 would be a positive value. If the value is negative this means the wound size has grown in size.
Time Frame: Baseline and four weeks
Population: The intention to treat population
Measure: Mean (95% Confidence Interval); unit: Percentage of wound area reduction
Arm/Group | Mepilex Border With Aquacel Extra Hydrofiber | Biatain® Silicone
Number analyzed (Participants) | 50 | 47
Percentage of wound area reduction | 43 [26.5 to 59.6] | 54.3 [37.1 to 71.5]

2. Secondary Outcome: Total Treatment Costs, £, During 4 Weeks Based on the Number of Dressings Used and the Unit Price in £ of the Products
Description: Total cost, £, was calculated as the number of products used multiplied by the unit price of the product. The price was extracted from the Drug Tariff on the date of Last Patient Out.
Time Frame: Baseline to 4 weeks
Population: Intention to treat population
Measure: Mean (95% Confidence Interval); unit: mean £
Arm/Group | Mepilex Border With Aquacel Extra Hydrofiber | Biatain® Silicone
Number analyzed (Participants) | 50 | 47
mean £ | 21.4 [16.9 to 26] | 14.3 [9.6 to 19]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study period, i.e., 4 weeks.
Arm/Group | Mepilex Border With Aquacel Extra Hydrofiber | Biatain® Silicone
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/51
Serious Adverse Events (participants affected / at risk) | 1/51 | 1/50
Other Adverse Events (participants affected / at risk) | 6/51 | 4/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Border With Aquacel Extra Hydrofiber (N=51) | Biatain® Silicone (N=50)
distended abdomen (Gastrointestinal disorders) | 1 (1) | 0 — Unlikely device related
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 — unlikely related to device
pulmonary embolism and atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Death due to suspected pulmonary embolism and atrial fibrillation. Unrelated to device
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Border With Aquacel Extra Hydrofiber (N=51) | Biatain® Silicone (N=50)
skin rash (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT05786612/Prot_SAP_000.pdf